CLINICAL TRIAL: NCT02760069
Title: Nasally Inhaled Isopropyl Alcohol Versus Oral Ondansetron for the Treatment of Nausea in the Emergency Department: A Double-Blind Randomized Controlled Trial
Brief Title: Isopropyl Alcohol vs Ondansetron for Nausea in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2016.091
Record Dates: First submitted 2016-04-15; First posted 2016-05-03 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — Ethanol; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inhaled ISO + oral ondansetron (Active Comparator): Inhaled isopropyl alcohol pads as needed for nausea (up to q30 minutes) and drink oral elixir comprising ondansetron (4 mg).
  Interventions: Drug: Inhaled isopropyl alcohol; Drug: Oral ondansetron
- Inhaled ISO + oral placebo (Experimental): Inhaled isopropyl alcohol pads as needed for nausea (up to q30 minutes) and drink oral placebo elixir.
  Interventions: Drug: Inhaled isopropyl alcohol; Drug: Oral placebo
- Inhaled placebo + oral ondansetron (Active Comparator): Inhaled normal saline pads as needed for nausea (up to q30 minutes) and drink oral placebo elixir.
  Interventions: Drug: Oral ondansetron; Drug: Inhaled normal saline

INTERVENTIONS:
Drug: Inhaled isopropyl alcohol — Patients will inhale from isopropyl alcohol pads as needed for nausea up to q30 minutes.
  Other Names: ISO
  Arms: Inhaled ISO + oral ondansetron; Inhaled ISO + oral placebo
Drug: Oral ondansetron — Patients will drink elixir containing 4 mg ondansetron in 5 ml of solution. National Drug Code (NDC) 0054-0064-47.
  Other Names: Ondansetron
  Arms: Inhaled ISO + oral ondansetron; Inhaled placebo + oral ondansetron
Drug: Inhaled normal saline — Patients will inhale from normal saline pads as needed for nausea up to q30 minutes.
  Other Names: Inhaled placebo
  Arms: Inhaled placebo + oral ondansetron
Drug: Oral placebo — Subjects will drink solution comprised of 0.25 ml of Oral Sweet Sugar Free NDC 0574-0302-16 with 4.75 ml of sterile water for dilution NDC 0264-2101-00
  Other Names: Oral sugar water
  Arms: Inhaled ISO + oral placebo

SUMMARY:
This study will compare the efficacy of isopropyl alcohol and conventional anti-emetics with three study arms: (1) inhaled isopropyl alcohol plus oral ondansetron; (2) inhaled isopropyl alcohol plus oral placebo; (3) inhaled placebo plus oral ondansetron.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial to test the hypothesis that nasally-inhaled isopropyl alcohol (ISO) plus oral placebo has greater anti-emetic efficacy compared to oral ondansetron oral solution. By design, the study will be double-blinded insofar as neither investigators nor subjects will be notified of the identity of the substances they are inhaling or swallowing. The study will include a post-study survey to ascertain the extent to which blinding was achieved. Potential subjects are those presenting to the Emergency Department (ED) with nausea and/or vomiting. Investigators will recruit a convenience sample by approaching subjects at the time of initial triage and solicit nausea on a verbal numerical rating scale (VNRS) scored from 0-10 with those patients reporting scores of 3 or greater eligible for study. Informed consent will be obtained from each subject.

Subjects will be allocated to one of three arms: (1) inhaled isopropyl alcohol plus oral ondansetron; (2) inhaled isopropyl alcohol plus oral placebo; (3) inhaled placebo plus oral ondansetron. No subject will receive both inhaled and oral placebo; all subjects will be allocated to at least one therapeutic intervention for nausea. Both investigators and study subjects will be blinded to subject allocation.

Regarding the interventions, upon recruitment, patients will be administered an oral solution (placebo or ondansetron) by their treating nurse. A study team member will then instruct the subject to inhale one of the blinded prep pads, to hold the pad approximately 1 centimeter from their nares, and to take deep nasal inhalations as needed for nausea relief. The investigator will remain at arm's length from the patient at all times to avoid detecting prep pad scent. Additionally, investigators will also instruct subjects to avoid any behavior or actions during the study that would indicate which preparation pad is being used.

The investigators will record their findings on data collection forms. The primary outcome will be nausea as measured on a 10 cm visual analogue scale (VAS) at 30 minutes. Nausea measurements will also be collected at 10, 20, 40, 50, and 60 minutes, and then every hour up to 5 hours, then at disposition at which time the patient will provide one final nausea VAS score. The study team member will not be present in the patient's room during the intervals between these evaluations. At the time of each nausea measurement, patients will be offered another preparation pad (up to ten pads). Investigators will notify the patient's treating provider to prompt consideration for treatment with a rescue anti-emetic (such as metoclopramide or promethazine) if the patient vomits or if the patient requests an anti-emetic at any time. At the time of each nausea measurement, a pain score will also be measured on a 10 cm VAS. At the time of final disposition, the patient will provide a satisfaction score on a 10-cm VAS and be asked to indicate his/her belief as to whether the pad was a treatment or placebo and whether the oral solution was a treatment or placebo. Similarly, at study conclusion the patient's provider will be asked to indicate his/her belief as to whether the pad was a treatment or placebo and whether the oral solution was a treatment or placebo. Other data collected will include times and doses for all medications (including preparation pads) and fluids administered, episodes of vomiting (defined as forceful expulsion of gastric contents separated by at least 2 minutes), disposition (admission versus discharge), final clinical impression at the time of disposition, and time to disposition. Subjects will be followed and data collected for the entirety of their ED stay.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older
* complaint of nausea and/or vomiting reported at 3 or above on verbal numerical rating scale at the time of triage

Exclusion Criteria:

* allergy to isopropyl alcohol or ondansetron
* inability to breathe through nose (e.g., recent upper respiratory infection)
* intake of cefoperazone, disulfiram, or metronidazole within the last 24 hours
* mental status precluding informed consent including intoxication
* known QT-prolongation
* clinical suspicion for serotonin syndrome
* intravenous catheter in place prior to study start
* medications administered since patient arrival (e.g., in triage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D April, MD, PhD, MSc, Principal Investigator — Brooke Army Medical Center
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beadle KL, Helbling AR, Love SL, April MD, Hunter CJ. Isopropyl Alcohol Nasal Inhalation for Nausea in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):1-9.e1. doi: 10.1016/j.annemergmed.2015.09.031. Epub 2015 Dec 8. PMID 26679977
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD007598. doi: 10.1002/14651858.CD007598.pub2. PMID 22513952
- [Background] Egerton-Warburton D, Meek R, Mee MJ, Braitberg G. Antiemetic use for nausea and vomiting in adult emergency department patients: randomized controlled trial comparing ondansetron, metoclopramide, and placebo. Ann Emerg Med. 2014 Nov;64(5):526-532.e1. doi: 10.1016/j.annemergmed.2014.03.017. Epub 2014 May 10. PMID 24818542
- [Derived] April MD, Oliver JJ, Davis WT, Ong D, Simon EM, Ng PC, Hunter CJ. Aromatherapy Versus Oral Ondansetron for Antiemetic Therapy Among Adult Emergency Department Patients: A Randomized Controlled Trial. Ann Emerg Med. 2018 Aug;72(2):184-193. doi: 10.1016/j.annemergmed.2018.01.016. Epub 2018 Feb 17. PMID 29463461

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled ISO + Oral Ondansetron | Inhaled ISO + Oral Placebo | Inhaled Placebo + Oral Ondansetron
Started | 40 | 41 | 41
Completed | 40 | 40 | 40
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled ISO + Oral Ondansetron | Inhaled ISO + Oral Placebo | Inhaled Placebo + Oral Ondansetron | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 38 | 117
  >=65 years | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 21 | 55
  Male | 20 | 26 | 19 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 6 | 21
  White | 28 | 34 | 33 | 95
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120
Nausea 100-mm visual analogue scale [Mean (Standard Deviation); unit: units on a scale] — Full Scale Name: Nausea 100-mm visual analogue scale. Scale Construct: Measures nausea as reported by the patient Scale Range: Minimum is 0 (no nausea) to 100 (worst nausea imaginable). These values quantify, on an interval scale anchored at 0, the patient's subjective sensation of nausea. Higher values represent worse outcomes (e.g., more nausea). Patient makes a single vertical mark on a 100 mm horizontal line with 0 at the left and 100 on the right to depict their nausea.
  units on a scale | 53 (22) | 51 (21) | 51 (20) | 52 (21)

OUTCOME MEASURES:

1. Primary Outcome: Nausea 100 mm Visual Analogue Scale (VAS)
Description: Full Scale Name: Nausea 100-mm visual analogue scale. Scale Construct: Measures nausea as reported by the patient Scale Range: Minimum is 0 (no nausea) to 100 (worst nausea imaginable). These values quantify, on an interval scale anchored at 0, the patient's subjective sensation of nausea. Higher values represent worse outcomes (e.g., more nausea). Patient makes a single vertical mark on a 100 mm horizontal line with 0 at the left and 100 on the right to depict their nausea.
Time Frame: 30 minutes post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inhaled ISO + Oral Ondansetron | Inhaled ISO + Oral Placebo | Inhaled Placebo + Oral Ondansetron
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 23 (25) | 19 (18) | 42 (27)

2. Secondary Outcome: Number of Participants Who Required Rescue Anti-emetics
Description: Whether patient required rescue anti-emetics (binary variable). Measured using nurse drug administration record.
Time Frame: Study duration (up to 5 hours post intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled ISO + Oral Ondansetron | Inhaled ISO + Oral Placebo | Inhaled Placebo + Oral Ondansetron
Number analyzed (Participants) | 40 | 40 | 40
Participants | 11 | 10 | 18

ADVERSE EVENTS:
Time Frame: Duration of study (up to 5 hours)
Arm/Group | Inhaled ISO + Oral Ondansetron | Inhaled ISO + Oral Placebo | Inhaled Placebo + Oral Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT02760069/Prot_SAP_000.pdf